CLINICAL TRIAL: NCT05224453
Title: Comparative Effects of Integrated Physical Training With High Protein Diet Versus Low Protein Diet in COVID-19 Asymptomatic Older Adults With Sarcopenia Symptoms.
Brief Title: Integrated Physical Training With Protein Diet in Older Adults With Sarcopenia Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RHPT/020/051
Record Dates: First submitted 2022-01-20; First posted 2022-02-04 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Sarcopenia
Keywords: COVID-19; Sarcopenia; physical training; muscle strength; muscle mass; Quality of life; protein diet
MeSH Terms: conditions — Sarcopenia; COVID-19 | interventions — Diet, High-Protein; Diet, Protein-Restricted

STUDY DESIGN:
Intervention Model Description: Single-blinded, randomized, experimental study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical training and high protein diet (Other): Subjects in this group underwent integrated physical training for 8 weeks. In addition to the integrated physical training exercises, group A received a high protein diet in the range of 1.1 - 1.3 g/kg protein/ ideal body weight/day (>1 g/kg aBW/d).
  Interventions: Other: Physical training and high protein diet
- Physical training and low protein diet (Other): Subjects in this group underwent integrated physical training for 8 weeks. In addition to the integrated physical training exercises, group B received a low protein diet in the range of 0.7 - 0.9 g/kg protein/ ideal body weight/day (<1 g/kg aBW/d)
  Interventions: Other: Physical training and low protein diet

INTERVENTIONS:
Other: Physical training and high protein diet — In addition to the integrated physical training exercises, group A received a high protein diet in the range of 1.1 - 1.3 g/kg protein/ ideal body weight/day (>1 g/kg aBW/d)
  Arms: Physical training and high protein diet
Other: Physical training and low protein diet — In addition to the integrated physical training exercises, group B received low protein diet in the range of 0.7 - 0.9 g/kg protein/ ideal body weight/day (<1 g/kg aBW/d)
  Arms: Physical training and low protein diet

SUMMARY:
Sarcopenia is the major health concern and common consequence of COVID-19 in the aging population. Moreover, this clinical condition has not been considered in usual physical rehabilitation practice, and its optimal protein requirement in food is not well defined, which requires a meaningful study in this field. The reports of this trial would deliver the latest evidence and proper guidelines for the prescription of physical exercises and also provide an optimal dietary plan in sarcopenia patients with COVID infection.

Objective: To find and compare the clinical and psychological effects of integrated physical training with a high protein diet versus a low-protein diet in community-dwelling COVID-19 asymptomatic older adults with Sarcopenia symptoms.

DETAILED DESCRIPTION:
It is a single-blinded, randomized, experimental study performed from March -2020 to November-2021. The trial received acceptance from the department of the ethical committee (DEC), Prince Sattam bin Abdulaziz University, Al-Kharj, Saudi Arabia with an approval number of RHPT/020/51. The DEC approved the subject consent form, treatment protocols, and the outcome parameters measured in the trial. The trial was executed in accordance with the ethical guidelines laid down in the 1964 Declaration of Helsinki. The finally selected subjects for the trial were asked to fill out the written subject consent form and underwent measurements for pre-interventional personal and anthropometric data. A two-block simple random sampling method was used to randomize and allocated the participants into two treatment groups. Group A was treated with integrated physical training with a high protein diet (n = 38) and group B was treated with the same integrated physical training with a low protein diet (n = 38) for a duration of eight weeks.

Subjects' personal and anthropometric measurements were calculated through Kolmogorov-Smirnov test for testing homogeneity and the data were represented in tabular form. The measurements were taken before the intervention, during the intervention at 4 weeks, after intervention at 8 weeks and after 6 months follow up. The data were shown as mean and standard deviation with 95% confidence interval (CI) with upper and lower limits. The time and group (4 × 2) multiple analysis of variance (MANOVA) of primary and secondary variables are reported between group A and group B at various intervals. The student's t-test was used to calculate inter-group effects and repeated measures (rANOVA) were used to calculate the intra-group effects. IBMSPSS - online version 20 was used to do all the statistical tests and the α level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Sarcopenia was diagnosed according to the guidelines given by the Asian working group for Sarcopenia (AWGS).

Appendicular skeletal muscle mass index (ASMI< 7.0 kg/m2) Patients with less muscle mass, Low handgrip strength (< 24 kg) Decrease walking speed (< 0.7 m/sec)

Exclusion Criteria:

Subjects with a history of physical workout, Taking medicines Recent surgeries Joint problems in the leg Heart and lung problems Neurological issues Other systemic diseases Contraindications for physical training

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with 60 - 80 years of age
Enrollment: 76 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All the data can be obtained by contacting the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one week.
Access Criteria: IPD can be obtained by contacting principal investigator

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 01-03-2020 to 30-11-2021 at Department of Physical therapy, Prince Sattam bin Abdulaziz University, Al-Kharj, Saudi Arabia
Pre-assignment Details: The finally selected subjects for the trial were asked to fill out the written subject consent form and underwent measurements for pre-interventional personal and anthropometric data. Their baseline primary and secondary outcome measures were also measured.
Period: Overall Study
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
Started | 38 | 38
Completed | 36 | 35
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (3.8) | 64.5 (3.6) | 64.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 00 | 00 | 0
  Male | 38 | 38 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height (m) [Mean (Standard Deviation); unit: metre] | 1.64 (0.23) | 1.68 (0.25) | 1.66 (0.24)
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 78.8 (4.3) | 79.2 (3.8) | 79.0 (4.0)
BMI (kg/m^2 ) [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (1.8) | 23.4 (1.9) | 23.3 (1.85)
VO2peak (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] | 30.8 (1.9) | 31.1 (1.6) | 30.9 (1.7)
HR (beats/min) [Mean (Standard Deviation); unit: beats/min] | 78.1 (4.5) | 79.2 (4.6) | 78.6 (4.55)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Hand Grip Strength
Description: The test is easy to perform and a less expensive one. It measures the strength of upper extremity by using a device handheld dynamometer. The participant was instructed to press the hand piece of the dynamometer to the maximum of his ability and the values shown on the display were recorded. Three values were noted for each participant and the mean value was considered for interpretation and it is a reliable and valid tool to measure the strength of upper extremity.
Time Frame: At baseline and at 6 months
Population: At baseline and at 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
Number analyzed (Participants) | 36 | 35
kg
  At Baseline | 29.2 (2.5) | 29.5 (2.4)
  At 6 months | 35.3 (2.8) | 30.3 (2.5)
Statistical Analysis 1: Comparison: Physical Training and High Protein Diet vs Physical Training and Low Protein Diet; Test type: Superiority — Parametric t test; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-6.21 to -3.78]

2. Secondary Outcome: Change in Muscle Cross Sectional Area
Description: Muscle CSA is measured with Magnetic resonance imaging (MRI) scan and it is an expensive measurement. The CSA of three major muscle such as;half way at arm - biceps, thigh - quadriceps and calf muscles were measured and included for analysis.
Time Frame: At baseline and at 6 months
Population: At baseline and at 6 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
Number analyzed (Participants) | 36 | 35
cm^2
  MRI - mid arm: At baseline | 54.9 (4.2) | 55.1 (4.3)
  MRI - mid arm: At 6 months | 58.9 (4.7) | 57.2 (4.7)
  MRI - mid thigh: At baseline | 65.2 (5.5) | 64.9 (5.4)
  MRI - mid thigh: At 6 months | 71.2 (6.4) | 67.5 (6.0)
  MRI - mid calf: At baseline | 61.8 (4.7) | 60.9 (4.6)
  MRI - mid calf: At 6 months | 67.2 (5.3) | 62.8 (5.2)
Statistical Analysis 1: Comparison: Physical Training and High Protein Diet vs Physical Training and Low Protein Diet; Test type: Superiority — Parametric t test; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-6.53 to -0.86]
Statistical Analysis 2: Comparison: Physical Training and High Protein Diet vs Physical Training and Low Protein Diet; Test type: Superiority — Parametric t test; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.84 to 0.44]

3. Secondary Outcome: Changes in Kinesiophobia
Description: Tampa scale of kinesiophobia questionnaire - Tampa scale of kinesiophobia questionnaire was administered to find the level of fear of movement of participants. The questionnaire has eleven items, which measures the mindset at various activities on a four-point Likert scale (1- Strongly disagree, 2 - Disagree, 3 - Agree, 4 - Strongly agree). The maximum score indicates a high level of fear whereas the minimum score indicates a low level of fear during activities, where 11-21 means no kinesiophobia, 22-27 mild kinesiophobia, 28-33 moderate kinesiophobia, and 34-44 means severe kinesiophobia.
Time Frame: At baseline and at 6 months
Population: At baseline and at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
Number analyzed (Participants) | 36 | 35
units on a scale
  At baseline | 32.5 (3.3) | 32.7 (3.4)
  At 6 months | 14.2 (1.6) | 22.3 (2.4)

4. Secondary Outcome: Changes in Quality of Life
Description: Sarcopenia quality of life (SarQol) questionnaire: The sarcopenia quality of life (SarQol) questionnaire was used to measure the subjects' wellbeing. The participants filled out the questionnaire themselves and it is a robust tool to measure Quality of life. The maximum score indicates a high level of quality of life, whereas the minimum score indicates a low level of quality of life. The total scoring indicates 0-20: worst health, 21-40: poor health; 41-60: fair 61-80: good, and 81-100, best health.
Time Frame: At baseline and at 6 months
Population: At 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
Number analyzed (Participants) | 36 | 35
units on a scale
  At baseline | 57.1 (5.9) | 58.0 (5.8)
  At 6 months | 68.2 (5.9) | 61.9 (6.1)

ADVERSE EVENTS:
Time Frame: 6 months follow-up.
Description: No adverse reactions were noted.
Arm/Group | Physical Training and High Protein Diet | Physical Training and Low Protein Diet
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05224453/Prot_SAP_ICF_000.pdf